CLINICAL TRIAL: NCT02572544
Title: Comparison of Objective and Subjective Changes Induced by Multiple Pinhole Glasses and Single Pinhole Glasses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, WonSoo Kim, Department of Ophthalmology, Chung-Ang University Hospital, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ChungAngUHeye
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Functional Vision Changes
Keywords: young healthy adults; single pinhole glasses; multiple pinhole glasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants (Experimental): All participants perform all exams under 3 conditions, that is baseline, single pinhole glasses, and multiple pinhole glasses
  Interventions: Device: Trayner Pinhole Glasses (Trayner Glasses, Ivybridge Devon, U.K.)

INTERVENTIONS:
Device: Trayner Pinhole Glasses (Trayner Glasses, Ivybridge Devon, U.K.) — Wearing multiple and single pinhole glasses

SUMMARY:
Purpose of this study is to compare the ocular functional changes including pupil size, visual acuity, depth of focus, accommodative amplitude, visual field, contrast sensitivity, and stereopsis induced by multiple and single pinhole glasses, in addition, to check reading speed and survey for ocular discomfort after using both pinhole glasses.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 and 45 years;
2. spherical equivalents (SE) within ± 6.0 diopters (D);
3. correctable distant and near visual acuity by glasses up to 20/20;
4. normal intraocular pressure with normal optic disc appearance;
5. normal ocular alignment.

Exclusion Criteria:

1. disturbance of accommodation due to any reasons such as an Adie's pupil, Parkinson's disease, a history of previous ocular surgery or trauma, and a history of systemic or topical medication that might affect accommodation;
2. corneal pathologic features;
3. glaucoma;
4. cataracts of grade II or greater by the Lens Opacities Classification System III (LOCS III);
5. vitreous and retinal abnormalities that might limit the accuracy of testing.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Distant visual acuity (logMAR) | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Distant visual acuity were measured using Snellen chart (Precision Vision, La Salle, IL, USA) at 4 m.
Photopic pupil size (baseline, mm) | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Pupil size under photopic conditions (85 cd/m2) was measured using a WASCA Analyzer (Carl Zeiss Meditec, Oberkochen, Germany).
Depth of focus | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Monocular DOF was checked with a 4-m Snellen chart under distance correction without cycloplegics.
Accommodative amplitude (Diopter) | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Near point of accommodation (NPA) was measured using Donder's push-up method.
Standard automated perimetry | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Visual field (VF) test was performed with a Humphrey Visual Field Analyzer (Carl Zeiss Meditec, Inc., Dublin, CA, USA) using the 30-2 Swedish interactive threshold algorithm.
Contrast sensitivity | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Monocular contrast sensitivity test was performed using a CSV-1000E Contrast Testing Instrument (VectorVision, Dayton, OH, USA) at 2.5-m distance under standard brightness (85 cd/m2)
Stereopsis (seconds of arc) | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Stereopsis was checked with the Randot Stereotest (Stereo Optical Co., Chicago, IL, USA).
Reading speed (letters per second) | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Reading speed was evaluated using the famous Korean traditional fairy tale book. This Korean book was printed black-and-white with 10-font size. The time taken to read designated 10 pages including 3985 letters was recorded, and then reading speed was calculated as letters per second (LPS).
Near visual acuity (logMAR) | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Near visual acuity using Logarithmic Visual Acuity Chart 2000 (Precision Vision, La Salle, IL, USA) at 40 cm.
Pupil size with the both pinhole glasses (mm) | Subjects performed this examination while wearing multiple and single pinhole glasses with one week apart in random order after baseline study.
  Pupil size with the both pinhole glasses using the ruler attached to the lateral rim of the glasses.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim WS, Park IK, Park YK, Chun YS. Comparison of Objective and Subjective Changes Induced by Multiple-Pinhole Glasses and Single-Pinhole Glasses. J Korean Med Sci. 2017 May;32(5):850-857. doi: 10.3346/jkms.2017.32.5.850. PMID 28378561